CLINICAL TRIAL: NCT05541328
Title: Comparison of Clinical Outcomes Among Patients Treated With Tisagenlecleucel in the JULIET Trial Versus a Real-world, Retrospective Cohort of Patients Treated With Standard of Care for Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Comparison of Clinical Outcomes Among Patients Treated With Tisagenlecleucel
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCTL019C2002
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tisagenlecleucel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Tisagenlecleucel therapy: The trial cohort is defined as the cohort of patients enrolled in JULIET who were assigned to receive tisagenlecleucel infusion
  Interventions: Other: Tisagenlecleucel
- Standard of care: The real-world cohort is defined as the cohort of patients derived from the FHRD receiving SOC as the third line of therapy or later

INTERVENTIONS:
Other: Tisagenlecleucel — The trial cohort is defined as the cohort of patients enrolled in JULIET who were assigned to receive tisagenlecleucel infusion
  Groups: Tisagenlecleucel therapy

SUMMARY:
This is a non-interventional, retrospective cohort study using the Flatiron Health Research Database (FHRD) and data from the single-arm phase II JULIET clinical trial (NCT02445248).

DETAILED DESCRIPTION:
JULIET is a single-arm, open-label, multi-center phase II study of tisagenlecleucel involving adult patients with r/r DLBCL who were ineligible for or had disease progression after autologous hematopoietic stem-cell transplantation.

Patients enrolled in JULIET will be referred to as the trial cohort in this study. Outcomes observed in the trial cohort will be compared against a cohort of patients receiving standard of care, defined as the real-world cohort in this study. The real-world cohort will be derived from the FHRD by applying relevant JULIET trial inclusion and exclusion criteria that are feasible to apply in the FHRD.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with Non-Hodgkin lymphoma (International Classification of Diseases 9th revision [ICD 9]: 200x, 202x or ICD 10th revision [ICD 10]: C82x, C83x, C84x, C85x, C86x, C88x, C96x), as captured in the structured data on or after January 1, 2011 AND at least two documented clinical visits in the Flatiron Health network on or after 01 January 2011.

AND has abstracted diagnosis date of DLBCL on or after January 1, 2011 AND received at least three lines of therapy AND received rituximab AND received anthracycline/anthracenedione AND has at least one 3L+ with prior exposure to rituximab and prior exposure to at least one anthracycline/anthracenedione AND at least 18 years old at index line start AND did not receive a clinical study drug in or prior to the earliest eligible 3L+ line (this represented Flatiron data delivered as part of the 3L + DLBCL Spotlight study) AND with at least 180 days of potential follow-up from index date to Flatiron data cutoff AND relapsed or refractory disease after ≥ 1 lines of therapy AND with ECOG performance status of 0-1 (or missing) within 30 days prior to the index date AND with adequate renal function defined as: serum creatinine of ≤ 1.5 x ULN or eGFR ≥ 60 mL/min/1.73 m2 (or missing) AND with adequate liver function defined as: ALT ≤ 5 x ULN and bilirubin ≤ 2.0 mg/dl (or missing) AND with adequate bone marrow reserve defined as: ANC > 1,000/mm3 and ALC ≥ 300/mm3 and platelets ≥ 50,000/mm3 and hemoglobin > 8.0 g/dl (or missing) AND confirmation of index line of therapy via abstraction.

Exclusion Criteria:

Exclude patients who received anti-CD19, CAR-T/gene therapy or allogenic stem cell transplant prior to index date AND exclude patients who received CAR-T/gene therapy except Yescarta, clinical study drug or autologous hematopoietic stem cell transplant as the index line of therapy AND exclude patients with CNS involvement on or prior to index date AND exclude HIV positive patients on or prior to index date AND exclude patients with myocardial infarction within 6 months prior to index date AND exclude patients with previous or concurrent malignancy on or prior to the index date AND exclude patients with evidence of pregnancy on or prior to index date AND exclude patients with T-cell rich/histiocyte rich large B-cell lymphoma (THRBCL), primary mediastinal B-cell lymphoma (PMBCL), EBV positive DLBCL, or Burkitt lymphoma

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with tisagenlecleucel in the JULIET trial versus a real-world, retrospective cohort of patients treated with standard of care for relapsed or refractory diffuse large B-cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS): ITT population | throughout the study, approximately 5 years
  To evaluate the efficacy of tisagenlecleucel therapy as compared to the current SOC as measured by overall survival (OS) among patients with r/r DLBCL and treated with at least two prior lines of systemic therapy.
Overall survival (OS): FAS population | throughout the study, approximately 5 years
  To evaluate the efficacy of tisagenlecleucel therapy as compared to the current SOC as measured by overall survival (OS) among patients with r/r DLBCL and treated with at least two prior lines of systemic therapy.

SECONDARY OUTCOMES:
Overall response rate (ORR): ITT population | throughout the study, approximately 5 years
  To evaluate the efficacy of tisagenlecleucel therapy as compared to the current SOC as measured by overall response rate (ORR), which includes complete response (CR) and partial response (PR), among patients with r/r DLBCL and treated with at least two prior lines of systemic therapy.
Overall response rate (ORR): FAS population | throughout the study, approximately 5 years
  To evaluate the efficacy of tisagenlecleucel therapy as compared to the current SOC as measured by overall response rate (ORR), which includes complete response (CR) and partial response (PR), among patients with r/r DLBCL and treated with at least two prior lines of systemic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States